CLINICAL TRIAL: NCT04013880
Title: A Phase IB/II Study to Evaluate the Safety, Tolerability, and Efficacy of ASTX727 and FT-2102 in IDH1-Mutated Myelodysplastic Syndrome or Acute Myeloid Leukemia
Brief Title: ASTX727 and FT-2102 in Treating IDH1-Mutated Recurrent/Refractory Myelodysplastic Syndrome or Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry); Forma Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Paul Ferrell, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC HEM 18165; NCI-2019-04103 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2019-07-05; First posted 2019-07-10 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Recurrent Myelodysplastic Syndrome; Refractory Acute Myeloid Leukemia; Refractory Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — decitabine and cedazuridine drug combination; olutasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ASTX727, FT-2102) (Experimental): Patients receive CDA inhibitor E7727/decitabine combination agent ASTX727 PO QD on days 1-5 and IDH-1 inhibitor FT-2102 PO QD or BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Drug: IDH-1 Inhibitor FT-2102

INTERVENTIONS:
Drug: CDA Inhibitor E7727/Decitabine Combination Agent ASTX727 — Given by mouth
  Other Names: ASTX727
Drug: IDH-1 Inhibitor FT-2102 — Given by mouth
  Other Names: FT 2102, FT-2102, IDH1-R132 Inhibitor FT-2102

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of FT-2102 when given together with ASTX727 in treating patients with IDH1-mutated myelodysplastic syndrome or acute myeloid leukemia that has come back (recurrent) or does not respond to treatment (refractory). ASTX727 is an oral deoxyribonucleic acid (DNA) methyltransferase (DNMT) inhibitor. DNA methylation is necessary for cell differentiation and development. Changes to the methylation profile can lead to DNA instability which can cause diseases like cancer. DNMT inhibitors target and inhibit these changes. FT-2102 is an isocitrate dehydrogenase 1 (IDH1) inhibitor. IDH1 is a type of protein involved in metabolism, or the process of providing the body's cells with energy. FT-2102 may stop the abnormal IDH1 protein and may reduce 2-HG levels in diseased cells to levels found in normal cells. Giving ASTX727 and FT-2102 may work better in treating patients with myelodysplastic syndrome or acute myeloid leukemia compared to ASTX727 and FT-2102 alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* To evaluate the safety of IDH-1 inhibitor FT-2102 (FT-2102) in combination with CDA inhibitor E7727/decitabine combination agent ASTX727 (ASTX727) in myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML) patients with IDH1 R132 mutations. (Phase Ib)
* To evaluate the response rate (overall response rate [ORR], complete response [CR], complete remission with partial hematologic recovery (CRh), complete remission with incomplete blood count recovery [CRi], morphologic leukemia-free state [MLFS], partial response [PR]) of the combination of ASTX727 and the IDH1-inhibitor, FT-2102 in subjects with myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML) with IDH1 R132 mutations. (Phase II)

SECONDARY OBJECTIVES:

* To confirm the phase II recommended dosing level of FT-2102 and ASTX727 in combination. (Phase Ib)
* To determine the pharmacokinetics of FT-2102 and ASTX727 in combination. (Phase Ib)
* To determine the reduction of bone marrow blasts. (Phase II)
* To determine the overall survival and event-free survival. (Phase II)
* To determine the levels of 2-HG in the blood and blood cells after treatment. (Phase II)
* To determine the relationship of 2-HG reduction to clinical response. (Phase II)

OUTLINE: This is a phase Ib, dose-escalation of IDH-1 inhibitor FT-2102 followed by a phase II study.

Patients receive CDA inhibitor E7727/decitabine combination agent ASTX727 orally (PO) once daily (QD) on days 1-5 and IDH-1 inhibitor FT-2102 PO QD or twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 12 months, and then periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Must voluntarily sign an informed consent document (ICF)
* Morphologically confirmed diagnosis of MDS (inclusive of MDS/MPN) or AML in accordance with World Health Organization (WHO) diagnostic criteria
* Phase Ib: Subjects may have

  * Relapsed/refractory AML or MDS or
  * Treatment naive AML
* Phase II Expansion: Subjects may have

  * Relapsed/refractory AML or MDS or
  * Treatment naive AML or
  * Treatment naive MDS
* For patients with MDS, must have a Revised International Prognostics Scoring System (IPSS-R) risk category of intermediate, high, or very high
* Confirmed IDH1 R132 mutation
* A bone marrow biopsy must be performed and tissue collected for entrance to the trial
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Life expectancy of at least 3 months in the assessment of the investigator
* Recovery from the non-hematologic toxic effects of prior treatment to grade =< 1, or baseline value according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.03 classification (excluding infertility, alopecia, or grade 1 neuropathy)
* Must have adequate hepatic and renal function as demonstrated by the following:

ALT (SGPT) and/or AST (SGOT) ≤ 3x upper limit of normal (ULN); Direct bilirubin ≤ 1.5 x ULN(or ≤ 2x ULN if due to Gilbert's disease); Serum creatinine of 1.5 x ULN or creatinine clearance of > 50 mL/min (whichever is lower)

* Baseline Fridericia's correction formula (QTcF) =< 450 msec (average of the QTcF values of screening triplicate electrocardiography [ECG]swith approximately two-minute intervals ) except for those patients with a bundle branch block (BBB)
* For fertile men and women, agreement to use effective contraceptive methods for the duration of study participation and 90 days after the last dose of study medication

Exclusion Criteria:

* Treatment naive patients who are suitable for and willing to receive intensive induction chemotherapy
* Patients with active, uncontrolled infection. Patients with infection under active treatment and controlled with antibiotics are eligible
* Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol
* Known history of human immunodeficiency virus (HIV), or known active hepatitis A, B, or C infection (hepatitis B carriers with normal liver function test [LFT]s and undetectable viral loads are allowed)
* Women who are pregnant or nursing
* Organ transplant recipients other than bone marrow transplant
* Autologous hematologic stem cell transplant within 3 months of study entry. Allogeneic hematologic stem cell transplant within 6 months. Grade II, or greater, active graft-versus- host disease
* Use of an investigational drug within 21 days or 5 half-lives (whichever is shorter) prior to the first dose of FT-2102/ASTX727. For investigational drugs for which 5 half-lives is less than 21 days, a minimum of 10 days between termination of the investigational drug and administration of FT-2102/ASTX727 is required
* Any major surgery, chemotherapy, or immunotherapy within the last 21 days (limited palliative radiation is allowed >= 2 weeks); concurrent hydroxyurea is allowed if less than or equal to 2 grams daily
* Ongoing immunosuppressive therapy including systemic corticosteroids (prednisone or equivalent =< 20 mg daily allowed as clinically warranted). Patients are allowed to use topical or inhaled corticosteroids
* Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol.
* Patients unable to swallow oral medications, or patients with gastrointestinal conditions (e.g., malabsorption, resection, etc.) deemed by the Investigator to jeopardize intestinal absorption
* Patients receiving intrathecal chemotherapy for active central nervous system (CNS) disease
* Patients who have exhibited allergic reactions to a previously administered IDH1 inhibitor
* Patients with acute promyelocytic leukemia (APL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (Phase Ib) | Up to 30 days
  Graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Response rate (Phase II) | Approximately 12 months
  calculated for each cohort, together with 95% confidence intervals based on exact binomial distributions.

SECONDARY OUTCOMES:
To confirm the phase II recommended dosing level (1b) | At 28 days
Pharmacokinetics parameters (1b) | Approximately 12 months
  analysis of plasma concentrations during the dose escalation phase of the study
Reduction of bone marrow blasts (phase II) | Approximately 12 months
Overall survival (Phase II) | Up to 2 years
  Time from randomization to death due to any cause
Event-Free Survival (Phase II) | Up to 2 years
  Time from start of treatment to event that treatment was intended to prevent or delay
Measure change in levels of 2-HG in the blood and blood cells after treatment (Phase II) | Up to 12 months
Compare 2-HG change to clinical response (Phase II) | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ferrell, MD, Principal Investigator — Vanderbilt Medical Center